CLINICAL TRIAL: NCT01219322
Title: Intravenous Bicarbonate Identifies the Correct Position of Intravenous Catheter
Brief Title: Intravenous Sodium Bicarbonate Verifies Intravenous Position of Catheters in Anesthetized Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ilan Keidan, director of pediatric anesthesiology and pain service, Sheba Medical center, Israel, Sheba Medical Center, Department of Anesthesiology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: SHEBA-09-7458-IK-CTIL
Record Dates: First submitted 2010-10-10; First posted 2010-10-13 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: General Anesthesia
Keywords: general endotracheal anesthesia; ASA I or II
MeSH Terms: interventions — Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous bicarbonate (Experimental): Intravenous bicarbonate(05meq/cc ) 50 cc will be injected.
  Interventions: Drug: Sodium bicarbonate
- Intravenous injection of 50 cc normal saline (Placebo Comparator): Injection of volume equivalent of normal saline to compare the establish the effect of same volume as the experimental drug
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Sodium bicarbonate — single use of sodium bicarbonate and sterile water for injection 1:1 concentration 50 cc
  Other Names: 8.4% w/v Sodium bicarbonate B Braun Melsungen, Germany.
  Arms: intravenous bicarbonate
Drug: normal saline — intravenous normal saline volume equivalent to sodium bicarbonate
  Arms: Intravenous injection of 50 cc normal saline

SUMMARY:
Extravasation is an unintentional injection or leakage of fluids in the perivascular or subcutaneous space. Extravasation can be associated with tissue injury with various level of severity and long term consequences. Currently the confirmation of intravenous location of the Intravenous (IV) catheter requires close observation of the insertion site with sufficient infiltration in the perivascular area to allow detection of swelling, discoloration and discomfort. Under Anesthesia direct observation is frequently prohibited. IV sodium bicarbonate (SB) is used frequently to treat different metabolic conditions and is known to cause a temporary elevation of exhaled carbon dioxide. This study aim is to evaluate the safety and efficacy of intravenous SB as a detector of intravenous placement of an IV line in anesthetized patients.

Patients and Methods: The study has three parts, in part 1, the safety of subcutaneous injection of sodium bicarbonate was evaluated in 6 rats. In each animal the macroscopic and microscopic effects were evaluated and a safe dilution was determined. In the second part of the study the investigators will evaluated the efficacy of IV diluted SB to detect the proper location of IV catheters. 20 adult patients age 20 to 50 years will be enrolled. Patients all under general anesthesia with standard controlled ventilation via endotracheal tube. The correct placement of IV catheter will be confirmed by easy aspiration of blood from newly placed IV catheter. In each patient a bolus of 50 cc of 0.5 meq/cc SB or volume equivalent of normal saline will be injected in random order. The data collection will include patient's demographics, the presence or absence of an increase in the expired end-tidal carbon dioxide, onset and peak changes of end-tidal carbon dioxide as well as the hemodynamic changes after each injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (American Society of Anesthesiologists [ASA] I or II) volunteers

Exclusion Criteria:

* respiratory disease
* active smoking
* cardiovascular disease
* renal disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
change in end-tidal carbon dioxide | 0.5-2 minutes
  intravenous bicarbonate injected intravenously will cause an increase in end-tidal carbon dioxide within minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel